CLINICAL TRIAL: NCT06137677
Title: Child Sweet and Savory Snack Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty with recruitment.
Sponsor: Penn State University (Other)
Responsible Party: Principal Investigator, Barbara J. Rolls, Professor of Nutritional Sciences, Penn State University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: ChildFood701
Record Dates: First submitted 2023-11-14; First posted 2023-11-18 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Eating Behavior
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sweet Snack (Experimental): A sweet food will be served as the snack
  Interventions: Other: Sweet Snack
- Savory Snack (Experimental): A savory food will be served as the snack
  Interventions: Other: Savory Snack

INTERVENTIONS:
Other: Sweet Snack — A sweet food will be served for the snack
  Arms: Sweet Snack
Other: Savory Snack — A savory food will be served for the snack
  Arms: Savory Snack

SUMMARY:
The purpose of this study is to determine how consumption of a snack food affects the hedonic ratings of that snack food compared to other foods. The results will have implications for guidance about the provision of snacks for preschool children and may help in identifying strategies for the prevention of obesity in children.

ELIGIBILITY:
Inclusion Criteria:

* Children who are enrolled in a scheduled classroom of the participating childcare centers
* Children who are between the ages of 4 and 6 years old at the time of enrollment

Exclusion Criteria:

* Children who are allergic to any of the foods served
* Children whose diets exclude any of the foods served
* Children who are absent from the childcare center on the acclimation day or both study days
* Children who are not able to complete study measures (e.g. only use the anchors or have low variability for their liking ratings)

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 14 (Actual)
Dates: Start 2024-02-05 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-05-15 (Actual)

PRIMARY OUTCOMES:
Change between interventions in liking of each test food | Study weeks 1 and 2
  Change between interventions in liking (before to after consumption) of the 5 test foods, measured using a visual analog scale (0-100 points).
Change between interventions in ranked preference of each test food from before to after consumption | Study weeks 1 and 2
  Change in ranked preference (before to after consumption) of the 5 test foods.

SECONDARY OUTCOMES:
Change between interventions of intake by weight | Study weeks 1 and 2
  Weight (grams) of food and water consumed
Change between interventions of intake by energy | Study weeks 1 and 2
  Energy (kilocalories) of food consumed
Change between interventions in fullness ratings from before to after consumption | Study weeks 1 and 2
  Change in fullness ratings (before to after consumption) measured using a 4-point scale ranging from empty to full.

CONTACTS AND LOCATIONS:
Locations (1):
- The Pennsylvania State University, University Park, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No